CLINICAL TRIAL: NCT03397667
Title: The Aging Brain ANSWERS Program: Veterans Living With Alzheimer's and Traumatic Brain Injury and Caregiver Burden
Brief Title: The Aging Brain ANSWERS Program
Acronym: ABC ANSWERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Richard L. Roudebush VA Medical Center (U.S. Federal Agency); Cleveland State University (Other)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Scientist, Indiana University Center for Aging Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #1706902669; AZ160032 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-08-08; First posted 2018-01-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Alzheimer Disease; Veterans; Family Caregivers; Caregiver Burden; Quality of Life
MeSH Terms: conditions — Brain Injuries, Traumatic; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is blinded to which arm a dyad is enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Primary Care
  Interventions: Other: Control
- Intervention (Experimental): Primary Care plus ABC ANSWERS intervention
  Interventions: Other: ABC ANSWERS

INTERVENTIONS:
Other: ABC ANSWERS — Primary Care plus ABC ANSWERS
  Arms: Intervention
Other: Control — Primary Care as usual
  Arms: Control

SUMMARY:
This study will test the effectiveness of an intervention for Veterans diagnosed with Alzheimer's Disease (AD) or Traumatic Brain Injury (TBI) and the burden on their informal (family/friend) caregiver.

DETAILED DESCRIPTION:
The majority of people with Alzheimer's (AD) and Traumatic brain Injury (TBI) are cared for in primary care settings and receive significant amounts of care and assistance in activities of daily living from family members or friends.

The ABC ANSWERS intervention will incorporate and integrate the common features of an evidence-based collaborative care model for brain care, while also attending to the implementation barriers of delivering care and skills to dyads of patients with AD and TBI and their family caregivers.

The study team will conduct a 1-year randomized control trial (RCT) designed to improve the Quality of Life (QoL) of Veterans with AD and TBI, and their family caregivers, and decrease their family caregivers' burden. The dyads in the intervention group will receive primary care plus ABC ANSWERS. The control group will receive primary care.

ELIGIBILITY:
Inclusion Criteria:

* Veterans: 1)Diagnosis of AD or TBI 2) Receives Primary Care from Veterans Administration Medical Center (VAMC)
* Caregivers: 1) Primary caregiver (family or friend) of a Veteran with AD or TBI 2) Plans to provide care for 1 year or longer
* Both: 1) Over 18 years of age 2) Speak and understand English 3) access to telephone

Exclusion Criteria:

* Veterans: 1) Resides in nursing home or long term care facility 2) currently receiving care in GRACE clinic 3) Enrolled in ANSWERS-VA research study
* Caregivers: 1) Does not consider him/herself a caregiver for Veteran 2) Serious medical illness limiting ability to participate
* Both: Unable to contact within 10 calls Age < 18 years Either caregiver or Veteran denies that they have AD or a TBI Either the caregiver or Veteran does not want to participate Not fluent in the English language Difficulty hearing or talking by telephone Has a terminal illness (e.g., cancer, end of life condition with decreased life expectancy, renal failure requiring dialysis) History of hospitalization for alcohol or drug abuse History of severe mental illness (e.g., suicidal tendencies, severe untreated depression or bipolar disorder, or schizophrenia) Prisoner or on house arrest

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Caregivers Quality of Life at 12 months | Baseline to 12 months
  Measure of quality of life using the 12 item Logsdon's Quality of Life scale. Items are scored on a scale from 0-3, "poor to excellent". The higher the score, the better the reporting of item.

SECONDARY OUTCOMES:
Change from baseline Veterans Quality of Life at 12 months | Baseline to 12 months
  Measure of quality of life using the 12 item Logsden's Quality of Life scale. Items are scored on a scale from 0-3, "poor to excellent". The higher the score, the better the reporting of item.
Change from baseline Caregiver Burden at 12 months | Baseline to 12 months
  Caregiver burden is measured using the Oberst Caregiver Burden Scale (OCBS). This is a valid 15 item questionnaire that rates 15 different types of caregiving tasks for informal caregivers based on perceived time and difficulty of the task. For each item the caregiver chooses a value from not difficult(0) to extremely difficult (5). Scores are averaged across 15 items of the time and difficulty subscales, thus achieving a score between 1 and 5 for each.
Change from baseline Veteran depression at 12 months | Baseline to 12 months
  Measure of Veteran depression using the Center for Epidemilogic Scale -Depression (CESD).This is a twenty item questionnaire comprising of six scales reflecting major facets of depression. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Change from baseline Caregiver depression at 12 months | Baseline to12 months
  Measure of Caregiver depression using the Center for Epidemilogic Scale -Depression (CESD).This is a twenty item questionnaire comprising of six scales reflecting major facets of depression. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Change from baseline Veteran anxiety at 12 months | Baseline to 12 months
  Measure of anxiety using the Generalized Anxiety Disorder Scale (GAD-7). This is a seven item anxiety scale with a total score from 0-21. Items are scored from "Not at all" (0) to "Nearly everyday" (3). The higher the score, the more often anxiety symptoms are endorsed.
Change from Caregiver anxiety at 12 months | Baseline to 12 months
  Measure of anxiety using the Generalized Anxiety Disorder Scale (GAD-7). This is a seven item anxiety scale with a total score from 0-21. Items are scored from "Not at all" (0) to "Nearly everyday" (3). The higher the score, the more often anxiety symptoms are endorsed.
Change from Caregiver dyadic strain at 12 months | Baseline to 12 months
  This is a 12 item scale ranging from strongly agree (3) to strongly disagree (0). The higher the score the more the respondent agrees or endorses relationship strain.

CONTACTS AND LOCATIONS:
Locations (1):
- Richard L. Roudebush VAMC, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carnahan JL, Judge KS, Daggy JK, Slaven JE, Coleman N, Fortier EL, Suelzer C, Fowler NR. Supporting caregivers of veterans with Alzheimer's disease and traumatic brain injury: study protocol for a randomized controlled trial. Trials. 2020 Apr 19;21(1):340. doi: 10.1186/s13063-020-4199-1. PMID 32306982